CLINICAL TRIAL: NCT03997539
Title: A Randomized, Multicenter, Phase II Open-label Study of the Efficacy and Safety of Pyrotinib + Vinorelbine vs. Treatment of Physician's Choice in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab-Based Therapy
Brief Title: A Study of Pyrotinib Plus Vinorelbine in Comparison With Treatment of Physician's Choice in Participants With HER2-positive Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, wang shusen, clinical professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-002
Record Dates: First submitted 2019-06-13; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pyrotinib 320mg + vinorelbine (Experimental): pyrotinib 320mg tablets administered daily by mouth, vinorelbine 80 mg/m2 weekly (following a first cycle at 60 mg/m2) administered OV on day 1 and day 8 of 21 day cycle. Treatment lasts for two cycles
  Interventions: Drug: Pyrotinib; Drug: vinorelbine
- pyrotinib 400mg + vinorelbine (Experimental): pyrotinib 400mg tablets administered daily by mouth, vinorelbine 80 mg/m2 weekly (following a first cycle at 60 mg/m2) administered OV on day 1 and day 8 of 21 day cycle. Treatment lasts for two cycles
  Interventions: Drug: Pyrotinib; Drug: vinorelbine
- Pyrotinib + vinorelbine (Experimental): pyrotinib administered daily by mouth（MTD）, vinorelbine 80 mg/m2 weekly (following a first cycle at 60 mg/m2) administered OV on day 1 and day 8 of 21 day cycle. Treatments will lasts until disease progression (as assessed by the investigator) or unmanageable toxicity.
  Interventions: Drug: Pyrotinib; Drug: vinorelbine
- Treatment of physician's choice (Active Comparator): Treatment of physician's choice until disease progression (as assessed by the investigator) or unmanageable toxicity. The treatments included single-agent chemotherapy, single-agent or dual-agent hormonal therapy for hormone receptor positive-disease, and single-agent HER2-directed therapy.
  Interventions: Drug: Treatment of physician's choice

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib Maleate combine with vinorelbine as the second-line treatment to HER2-positive Metastatic Breast Cancer
  Arms: Pyrotinib + vinorelbine; pyrotinib 320mg + vinorelbine; pyrotinib 400mg + vinorelbine
Drug: Treatment of physician's choice — The treatment of physician's choice (TPC) was a protocol-specified approved or standard of care therapy or combination of therapies, based on frequently used regimens for second-line HER2-positive metastatic breast cancer treatment after receipt of trastuzumab-containing regimens. The therapies included single-agent chemotherapy, single-agent (e.g., tamoxifen or aromatase inhibitor) or dual-agent (e.g., aromatase inhibitor with luteinizing hormone releasing hormone [LHRH] agonist) hormonal therapy for hormone receptor positive-disease, and single-agent HER2-directed therapy.
  Arms: Treatment of physician's choice
Drug: vinorelbine — vinorelbine
  Arms: Pyrotinib + vinorelbine; pyrotinib 320mg + vinorelbine; pyrotinib 400mg + vinorelbine

SUMMARY:
The purpose of this study is to identify the highest tolerable dose of pyrotinib in combination with vinorelbine and to assess the safety and efficacy of the combination in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer.

The study will be conducted in two parts. In the first part, testing will be done on up to 12 subjects to determine the highest tolerable dose of pyrotinib and vinorelbine in patients with advanced solid tumors. In the second part of the study, we will compare the safety and efficacy of Pyrotinib + vinorelbine vs. Treatment of Physician's Choice in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab-Based Therapy.Participants will be treated until disease progression (PD), unmanageable toxicity, or study termination.

ELIGIBILITY:
Inclusion Criteria:

* HER2 status must be prospectively, centrally tested and be HER2-positive based on central laboratory assay results
* Histologically or cytologically confirmed invasive breast cancer
* Prior treatment for breast cancer in the adjuvant, unresectable, locally advanced, or metastatic setting must include both a taxane, alone or in combination with another agent, and trastuzumab, alone or in combination with another agent
* Documented progression (which occur during or after most recent treatment or within 6 months after completing of adjuvant therapy) of incurable, unresectable, locally advanced or metastatic breast cancer, defined by the investigator
* Measurable and/or nonmeasurable disease; participants with central nervous system-only disease are excluded
* Cardiac ejection fraction greater than or equal to (>/=) 50 percent (%) by either echocardiogram or multi-gated acquisition scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* History of treatment with pyrotinib
* Prior treatment with lapatinib or neratinib
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma
* History of receiving any anti-cancer drug/biologic or investigational treatment within 28 days prior to randomization except hormone therapy
* Recovery of treatment-related toxicity consistent with other eligibility criteria
* History of radiation therapy within 28 days of randomization
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms, as well as any history of radiation, surgery, or other therapy, including steroids, to control symptoms from brain metastases within 2 months (60 days) of randomization
* History of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction or unstable angina
* Current severe, uncontrolled systemic disease (for example, clinically significant cardiovascular, pulmonary, or metabolic disease)
* Pregnancy or lactation
* Current known active infection with human immunodeficiency virus (HIV) or hepatitis C virus
* Presence of conditions that could affect gastrointestinal absorption: Malabsorption syndrome, resection of the small bowel or stomach, and ulcerative colitis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
maximum-tolerated dose (MTD) | 42 days
  The maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one subject out of three experiences has a dose-limiting toxicity (DLT) upon completing two treatment cycle.
PFS as Assessed by the Investigator | From enrollment to progression or death (for any reason),assessed up to 100 months
  progression-free survival

SECONDARY OUTCOMES:
Objective Response Rate | from enrollment to progression or death (for any reason), assessed up to 100 months
  CR+PR
OS | from enrollment to death (for any reason).assessed up to 100 months
  OS was defined as the time from the date of randomization to the date of death from any cause